CLINICAL TRIAL: NCT01917266
Title: Evaluation of Left Ventricular (LV) Lead Positioning Using MediGuide
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: SJM-CIP-10084
Record Dates: First submitted 2013-07-30; First posted 2013-08-06 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Concordant
- Discordant

SUMMARY:
The purpose of this study is to evaluate Cardiac Resynchronization Therapy(CRT) response in subjects with concordant versus discordant left ventricular (LV) lead position as compared to the site of latest mechanical activation.

ELIGIBILITY:
Inclusion Criteria:

* Be scheduled to undergo implant of a Cardiac Resynchronization Therapy (CRT) system with approved standard indication per accepted guidelines as a new implant or an upgrade from an existing Implantable Cardioverter Defibrillator (ICD) or pacemaker with no prior left ventricular lead placement
* Be in sinus rhythm at the time of enrollment
* Have the ability to provide informed consent for study participation and be willing and able to comply with the Clinical Investigational Plan described evaluations

Exclusion Criteria:

* Have persistent or permanent atrial fibrillation
* Be in New York Heart Association (NYHA) IV functional class
* Have prior left ventricular (LV) lead implant
* Be pacemaker-dependent
* Have a recent myocardial infarction within 40 days prior to enrollment
* Have undergone cardiac bypass surgery or coronary revascularization procedure within 3 months prior to enrollment or be scheduled for such procedures in the following 7 months
* Have had a recent Cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 3 months prior to enrollment
* Have had intravenous inotropic support in the last 30 days
* Exhibit Cheyne-Stokes respiration
* Be less than 18 years of age
* Be pregnant or planning to become pregnant during the duration of the investigation
* Be currently participating in any other clinical investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients indicated for a Cardiac Resynchronization Therapy (CRT) device
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Percent of patients with the left ventricle (LV) lead implanted at the site of latest mechanical activation | This outcome measure will be assessed after an off-line analysis immediately after implant

SECONDARY OUTCOMES:
Response to Cardiac Resynchronization Therapy (CRT) as defined by percent change in end-systolic volume (ESV) at 6-month follow-up relative to baseline. | 6 months after implant

CONTACTS AND LOCATIONS:
Locations (1):
- Herzzentrum Leipzig GmbH, Leipzig, Germany